CLINICAL TRIAL: NCT01142726
Title: A Phase 3b, Randomized, Active Controlled Trial to Evaluate the Efficacy and Safety of Abatacept SC in Combination With Methotrexate in Inducing Clinical Remission Compared to Methotrexate Monotherapy in Adults With Very Early RA
Brief Title: Efficacy and Safety Study of Abatacept Subcutaneous Plus Methotrexate in Inducing Remission in Adults With Very Early Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-226; 2010-018674-20 (EudraCT Number)
Record Dates: First submitted 2010-06-03; First posted 2010-06-11 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Abatacept, 125 mg, plus methotrexate, 2.5 mg (Active Comparator): Participants received abatacept, 125 mg subcutaneously, plus methotrexate, 2.5 mg orally as tablets, once weekly, during the 12-month Treatment Period
  Interventions: Drug: Abatacept; Drug: Methotrexate
- Methotrexate, 2.5 mg, plus abatacept placebo (Active Comparator): Participants received methotrexate, 2.5 mg, orally as tablets, plus abatacept placebo subcutaneously, once weekly during the 12-month Treatment Period
  Interventions: Drug: Methotrexate; Drug: Abatacept placebo
- Abatacept, 125 mg, plus methotrexate placebo (Active Comparator): Participants received abatacept, 125 mg subcutaneously, plus methotrexate placebo tablets orally, once weekly during the 12-month Treatment Period
  Interventions: Drug: Abatacept; Drug: Methotrexate placebo

INTERVENTIONS:
Drug: Abatacept — Injection, subcutaneous, 125 mg by syringe, once weekly, 12 months
  Other Names: Orencia; BMS 188667
  Arms: Abatacept, 125 mg, plus methotrexate placebo; Abatacept, 125 mg, plus methotrexate, 2.5 mg
Drug: Methotrexate — Tablets, oral, 2.5 mg, once weekly, 12 months
  Other Names: Rheumatrex
  Arms: Abatacept, 125 mg, plus methotrexate, 2.5 mg; Methotrexate, 2.5 mg, plus abatacept placebo
Drug: Abatacept placebo — Injection, subcutaneous, to match 125 mg by syringe, once weekly, 12 months
  Arms: Methotrexate, 2.5 mg, plus abatacept placebo
Drug: Methotrexate placebo — Tablets, oral, to match 2.5-mg tablet, once weekly, 12 months
  Arms: Abatacept, 125 mg, plus methotrexate placebo

SUMMARY:
The primary purpose of the protocol is to demonstrate the ability of abatacept plus methotrexate to induce remission in patients with very early rheumatoid arthritis after 12 months of treatment and to maintain remission following 6 months of drug withdrawal.

ELIGIBILITY:
Key Inclusion Criteria:

* Presence of active clinical synovitis in at least 2 joints, 1 of which must have been a small joint, for a minimum of 8 weeks prior to screening
* Onset of persistent symptoms ≤ 2 years prior to screening
* Positive test result for anticyclic citrullinated peptides 2
* Methotrexate naive or with minimum exposure to methotrexate, defined as no more than 10 mg/week for ≤4 weeks and no methotrexate dose for 1 month prior to screening visit
* Biologic naive, including no treatment with an investigational biologic prior to screening
* Disease Activity Score 28 based on C-reactive protein score ≥3.2 at screening
* Withdrawal from any treatment with chloroquine, hydroxychloroquine, and/or sulfasalazine (wash-out) for a minimum of 28 days prior to randomization
* If receiving oral corticosteroids, on a stable low dose (≤ 10 mg/day prednisone equivalent) for at least 4 weeks
* Able to undergo magnetic resonance imaging

Key Exclusion Criteria:

* Meeting diagnostic criteria for other rheumatic disease (eg, lupus erythematosus)
* Treatment with an intravenous, intramuscular, or intraarticular corticosteroid within 4 weeks prior to randomization
* Scheduled for or anticipating joint replacement surgery
* Presence of concomitant illness likely to require systemic glucocorticosteroid therapy during the study, in the opinion of the investigator
* History of malignancy in the last 5 years
* Any serious bacterial infection within the last 3 months not treated or resolved with antibiotics, or any chronic or recurrent bacterial infection
* At risk for tuberculosis
* Evidence of active or latent bacterial or viral infection at the time of potential enrollment, including human immunodeficiency or herpes zoster virus or cytomegalovirus that resolved less than 2 months prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2010-12; Primary Completion 2013-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (64):
- United States (15):
  - Rheumatology Associates Of North Alabama, P.C., Huntsville, Alabama
  - St. Joseph'S Mercy Clinic, Hot Springs, Arkansas
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Coeur D'Alene Arthrit Clin, Coeur d'Alene, Idaho
  - Johns Hopkins University Division Of Rheumatology, Baltimore, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Arthritis Associates Of Mississippi, Jackson, Mississippi
  - Physician Research Collaboration, Llc, Lincoln, Nebraska
  - Piedmont Rheumatology, Pa, Hickory, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - Metrohealth Medical Center, Cleveland, Ohio
  - Isam A. Diab, Md, Middleburg, Ohio
  - Alan J. Kivitz, Md, Cpi, Duncansville, Pennsylvania
  - Mitchell C. Feinman, Md, Orangeburg, South Carolina
  - Kurt Oelke, Md, Glendale, Wisconsin
- Australia (6):
  - Local Institution, Cairns, Queensland
  - Local Institution, Maroochydore, Queensland
  - Local Institution, Woodville, South Australia
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Malvern, Victoria
  - Local Institution, Victoria Park, Western Australia
- Belgium (3):
  - Local Institution, Brussels
  - Local Institution, Kortrijk
  - Local Institution, Merksem
- Canada (2):
  - Local Institution, Calgary, Alberta
  - Local Institution, Laval, Quebec
- Local Institution, Hjørring, Denmark
- Finland (2):
  - Local Institution, Helsinki
  - Local Institution, Tampere
- France (4):
  - Local Institution, Chambray-lès-Tours
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Poitiers
- Germany (3):
  - Local Institution, Berlin
  - Local Institution, Hildesheim
  - Local Institution, München
- Italy (2):
  - Local Institution, Ancona
  - Local Institution, Siena
- Mexico (7):
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, San Luis Potosí City, San Luis Potosí
  - Local Institution, Metepec, State of Mexico
  - Local Institution, Mérida, Yucatán
  - Local Institution, Querétaro
- Poland (5):
  - Local Institution, Lublin
  - Local Institution, Poznan
  - Local Institution, Torun
  - Local Institution, Warsaw
  - Local Institution, Wroc#aw
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Tver'
- South Africa (4):
  - Local Institution, Kempton Park, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Panorama, Western Cape
- South Korea (3):
  - Local Institution, Daegu
  - Local Institution, Daejeon
  - Local Institution, Seoul
- Sweden (5):
  - Local Institution, Gothenburg
  - Local Institution, Linköping
  - Local Institution, Malmo
  - Local Institution, Stockholm
  - Local Institution, Uppsala

REFERENCES:
- [Derived] Ahmad HA, Baker JF, Conaghan PG, Emery P, Huizinga TWJ, Elbez Y, Banerjee S, Ostergaard M. Prediction of flare following remission and treatment withdrawal in early rheumatoid arthritis: post hoc analysis of a phase IIIb trial with abatacept. Arthritis Res Ther. 2022 Feb 16;24(1):47. doi: 10.1186/s13075-022-02735-8. PMID 35172859
- [Derived] Keystone EC, Ahmad HA, Yazici Y, Bergman MJ. Disease activity measures at baseline predict structural damage progression: data from the randomized, controlled AMPLE and AVERT trials. Rheumatology (Oxford). 2020 Aug 1;59(8):2090-2098. doi: 10.1093/rheumatology/kez455. PMID 31819995
- [Derived] Ahmad HA, Baker JF, Ostergaard M, Ye J, Emery P, Conaghan PG. Determining MRI Inflammation Targets When Considering a Rheumatoid Arthritis Treat-to-Target Strategy: Results of a Randomized, Placebo-Controlled Trial. Adv Ther. 2019 Sep;36(9):2384-2393. doi: 10.1007/s12325-019-01020-6. Epub 2019 Jul 5. PMID 31278695
- [Derived] Emery P, Burmester GR, Bykerk VP, Combe BG, Furst DE, Maldonado MA, Huizinga TW. Re-treatment with abatacept plus methotrexate for disease flare after complete treatment withdrawal in patients with early rheumatoid arthritis: 2-year results from the AVERT study. RMD Open. 2019 Feb 8;5(1):e000840. doi: 10.1136/rmdopen-2018-000840. eCollection 2019. PMID 30997151
- [Derived] Bykerk VP, Burmester GR, Combe BG, Furst DE, Huizinga TWJ, Ahmad HA, Emery P. On-drug and drug-free remission by baseline symptom duration: abatacept with methotrexate in patients with early rheumatoid arthritis. Rheumatol Int. 2018 Dec;38(12):2225-2231. doi: 10.1007/s00296-018-4173-3. Epub 2018 Oct 20. PMID 30341453
- [Derived] Peterfy C, Burmester GR, Bykerk VP, Combe BG, DiCarlo JC, Furst DE, Huizinga TW, Wong DA, Conaghan PG, Emery P. Sustained improvements in MRI outcomes with abatacept following the withdrawal of all treatments in patients with early, progressive rheumatoid arthritis. Ann Rheum Dis. 2016 Aug;75(8):1501-5. doi: 10.1136/annrheumdis-2015-208258. Epub 2016 Feb 10. PMID 26865601
- [Derived] Emery P, Burmester GR, Bykerk VP, Combe BG, Furst DE, Barre E, Karyekar CS, Wong DA, Huizinga TW. Evaluating drug-free remission with abatacept in early rheumatoid arthritis: results from the phase 3b, multicentre, randomised, active-controlled AVERT study of 24 months, with a 12-month, double-blind treatment period. Ann Rheum Dis. 2015 Jan;74(1):19-26. doi: 10.1136/annrheumdis-2014-206106. Epub 2014 Nov 3. PMID 25367713
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 511 patients were enrolled in the study, and 351 were randomized. The primary reasons that 160 enrolled patients were not randomized were failure to meet study criteria (130/160) and withdrawal of consent (20/160).
Groups:
- Abatacept, 125 mg, Plus Methotrexate, 2.5 mg: Participants received abatacept, 125 mg subcutaneously, plus methotrexate (MTX), 2.5 mg orally as tablets, once weekly, during the 12-month Treatment Period. Participants with a Low Disease Activity Score (LDAS) defined as DAS28-CRP score of < 3.2 at Month 12 (end of Treatment Period) entered the Withdrawal Period for up to 12 months, during which all study medication was withdrawn. Participants with a DAS28-CRP score of >3.2 were discontinued from the study. All MTX and corticosteroids, if not already discontinued, were to be tapered off during the first month of the Withdrawal Period. Participants who experienced a worsening of rheumatoid arthritis (RA) symptoms or a RA flare after at least 3 months in the Withdrawal Period were eligible to enroll into a 6-month Re-exposure Period, during which they received open-label treatment with abatacept subcutaneous (SC) 125 mg/week and MTX.
- Abatacept, 125 mg, Plus Methotrexate Placebo: Participants received abatacept, 125 mg subcutaneously, plus methotrexate placebo tablets orally, once weekly during the 12-month Treatment Period. Participants with a Low Disease Activity Score (LDAS) defined as DAS28-CRP score of < 3.2 at Month 12 (end of Treatment Period) entered the Withdrawal Period for up to 12 months, during which all study medication was withdrawn. Participants with a DAS28-CRP score of >3.2 were discontinued from the study. Participants who experienced a worsening of rheumatoid arthritis (RA) symptoms or a RA flare after at least 3 months in the Withdrawal Period were eligible to enroll into a 6-month Re-exposure Period, during which they received open-label treatment with abatacept SC (125 mg/week) and MTX.
- Methotrexate, 2.5 mg, Plus Abatacept Placebo: Participants received methotrexate, 2.5 mg, orally as tablets, plus abatacept placebo subcutaneously, once weekly during the 12-month Treatment Period. Participants with a Low Disease Activity Score (LDAS) defined as DAS28-CRP score of < 3.2 at Month 12 (end of Treatment Period) entered the Withdrawal Period for up to 12 months, during which all study medication was withdrawn. Participants with a DAS28-CRP score of >3.2 were discontinued from the study. All MTX and corticosteroids, if not already discontinued, were to be tapered off during the first month of the Withdrawal Period. Participants who experienced a worsening of rheumatoid arthritis (RA) symptoms or a RA flare after at least 3 months in the Withdrawal Period were eligible to enroll into a 6-month Re-exposure Period, during which they received open-label treatment with abatacept SC (125 mg/week) and MTX.
Period: Treatment Phase: Day 1 Through Month 12
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Started | 119 | 116 | 116
Completed | 103 | 91 | 96
Not Completed | 16 | 25 | 20
Not completed — Adverse Event | 5 | 8 | 5
Not completed — Withdrawal by Subject | 4 | 9 | 3
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Poor compliance/noncompliance | 1 | 0 | 0
Not completed — Lack of Efficacy | 5 | 6 | 11
Period: Withdrawal Phase: Months 12 up to 24
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Started | 84 | 66 | 75
Completed | 14 | 10 | 17
Not Completed | 70 | 56 | 58
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Pregnancy | 1 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — No longer met study criteria | 1 | 0 | 0
Not completed — Lack of Efficacy | 65 | 54 | 53
Not completed — non-specified | 0 | 1 | 1
Period: Re-Exposure Phase: Months 24 up to 30
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Started | 55 | 48 | 43
Completed | 54 | 46 | 40
Not Completed | 1 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients who received at least 1 dose of double-blind study medication in the Treatment Period
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo | Total
Number analyzed (Participants) | 119 | 116 | 116 | 351
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (13.20) | 45.4 (11.92) | 49.1 (12.36) | 47.0 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 89 | 89 | 273
  Male | 24 | 27 | 27 | 78
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 100 | 95 | 102 | 297
  Asian | 14 | 13 | 9 | 36
  Black/African American | 2 | 4 | 2 | 8
  American Indian/Alaska native | 1 | 1 | 1 | 3
  Other | 2 | 3 | 2 | 7
Duration of rheumatoid arthritis [Mean (Standard Deviation); unit: Years] | 0.58 (0.500) | 0.59 (0.522) | 0.50 (0.488) | 0.56 (0.504)
Disease Activity Score 28 based on C-reactive protein (DAS28-CRP) [Mean (Standard Deviation); unit: Units on a scale] — The DAS28-CRP is a measure of disease activity in rheumatoid arthritis (RA) and assesses the 28 joints RA commonly affects; the score includes the number of tender and swollen joints (out of 28), CRP level (a measure of inflammation in the blood), and the patient's global assessment of health (ranging from very good to very bad). These measures are then fed into a complex mathematical formula to produce the overall DAS (a score greater than 5.1 implies active disease; less than 3.2, well controlled disease; and less than 2.6, remission.)
  Units on a scale | 5.528 (1.2501) | 5.463 (1.1493) | 5.315 (1.3330) | 5.435 (1.2465)
Health Assessment Questionnaire Disability Index (HAQ-DI) score [Mean (Standard Deviation); unit: Units on a scale] — The HAQ-DI assesses patients' functional ability by rating their abilities over the previous week. It includes at least 2 questions from each of 8 categories: dressing and grooming, hygiene, arising, reach, eating, grip, walking, and common daily activities. Patients rate difficulty performing specific tasks: 0=without difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The sum of the categories score (the highest scored item in the category) is divided by the number of categories answered, yielding a score from 0-3.
  Units on a scale | 1.452 (0.6778) | 1.419 (0.6587) | 1.383 (0.6493) | 1.419 (0.6609)
Rheumatoid factor status [Number; unit: Participants]
  Positive | 113 | 111 | 110 | 334
  Negative | 6 | 5 | 6 | 17
Tender joint count [Mean (Standard Deviation); unit: Joints] | 24.3 (15.74) | 23.9 (14.47) | 21.7 (14.00) | 23.3 (14.77)
Swollen joint count [Mean (Standard Deviation); unit: Joints] | 16.5 (12.43) | 17.2 (12.88) | 15.7 (11.78) | 16.5 (12.35)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Remission by Disease Activity Score 28 Based on C-reactive Protein (DAS28-CRP) Criteria at Month 12 and at Both Months 12 and 18
Description: DAS28-CRP remission defined as <2.6; TP=treatment phase; WP=withdrawal phase. The DAS 28-CRP is a measure of disease activity in rheumatoid arthritis (RA) that assesses the 28 joints RA commonly affects; the score includes the number of tender and swollen joints (out of 28), CRP level (a measure of inflammation in the blood), and the patient's global assessment of health (ranging from very good to very bad). These measures are then fed into a complex mathematical formula to produce the overall DAS (a score greater than 5.1 implies active disease; less than 3.2, well controlled disease; and less than 2.6, remission.)
Time Frame: Randomization to Months 12 and 18
Population: All randomized participants who received at least 1 dose of double-blind study medication in the Treatment Period. Percentage calculated as a/b, where a=number of patients who achieved remission at Month 12 and at both Months 12 and 18, and b=number of patients in the analysis. n=number evaluable
Measure: Number; unit: Percentage of participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116
Percentage of participants
  Month 12 (TP Day 365) (n=115, 115) | 60.9 | 45.2
  Both Months 12 & 18 (WP Day 169) (n=115, 115) | 14.8 | 7.8
Statistical Analysis 1: Comparison: Abatacept, 125 mg, Plus Methotrexate, 2.5 mg vs Methotrexate, 2.5 mg, Plus Abatacept Placebo; Power estimate assumed 2-sided alpha level of 5% and that 60% of abatacept (ABA)+methotrexate (MX) patients (pts) would be in DAS28-CRP remission at Month 12 compared with 38% of MX monotherapy pts. Also assumed that 48% of ABA monotherapy pts would be in DAS28-CRP remission at Month 12, yielding an expected treatment difference from MX of 10% in favor of ABA monotherapy; 116 pts randomized to ABA monotherapy would yield a half-length of the 95% CI around that 10% treatment difference of 13.5%; Test type: Superiority or Other; p = 0.010, Regression, Logistic; Statistical testing of the 2 coprimary efficacy endpoints was conducted in a hierarchical fashion to maintain the overall Type I error rate at 5%; Odds Ratio (OR) = 2.01, 95% CI 2-sided [1.18 to 3.43], Standard Error of Mean 0.55 — At Month 12
Statistical Analysis 2: Comparison: Abatacept, 125 mg, Plus Methotrexate, 2.5 mg vs Methotrexate, 2.5 mg, Plus Abatacept Placebo; Conditional on statistical significance of the 1st coprimary efficacy analysis (CEA), a sample of 116 patients per arm would provide 98% power for the 2nd CEA comparison of the percentage of patients in DAS28-CRP remission at Months 12 and 18 between the abatacept (ABA)+methotrexate (MTX) arm and the MTX monotherapy arm for intent-to treat population. This sample size calculation assumed 30% remission in the ABA+MTX arm and 8% in the monotherapy arm at Month 18 and a 2-sided alpha level of 5%; Test type: Superiority or Other; p = 0.045, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.51, 95% CI 2-sided [1.02 to 6.18], Standard Error of Mean 1.15 — At Months 12 and 18

2. Secondary Outcome: Percentage of Participants Who Received Monotherapy and Achieved Remission by Disease Activity Score 28 Based on C-reactive Protein (DAS28-CRP) Criteria at Month 12 and at Both Months 12 and 18
Description: TP=treatment period; WP=withdrawal period. Remission defined as DAS28-CRP<2.6. The DAS 28-CRP is a measure of disease activity in rheumatoid arthritis (RA) that assesses the 28 joints RA commonly affects; the score includes the number of tender and swollen joints (out of 28), CRP level (a measure of inflammation in the blood), and the patient's global assessment of health (ranging from very good to very bad). DAS-CRP scores range from 0 to 10, with higher values indicating greater disease activity. Individual measures are fed into a complex mathematical formula to produce the overall DAS (a score greater than 5.1 implies active disease; less than 3.2, well controlled disease; and less than 2.6, remission.)
Time Frame: Randomization to Months 12 and 18
Population: All randomized participants who received at least 1 dose of double-blind monotherapy in the Treatment Period. Percentage calculated as a/b, where a=number of patients who achieved remission at Month 12 and at both Months 12 and 18, and b=number of patients in the analysis. n=number evaluable
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 116 | 116
Percentage of participants
  At Month 12 (TP Day 365) (n=113, 115) | 42.5 [33.36 to 51.59] | 45.2 [36.12 to 54.31]
  At both Months 12 &18 (WP Day 169) (n=113, 115) | 12.4 [6.31 to 18.46] | 7.8 [2.92 to 12.73]
Statistical Analysis 1: Comparison: Abatacept, 125 mg, Plus Methotrexate Placebo vs Methotrexate, 2.5 mg, Plus Abatacept Placebo; Test type: Superiority or Other; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.55 to 1.57], Standard Error of Mean 0.25 — At Month 12
Statistical Analysis 2: Comparison: Abatacept, 125 mg, Plus Methotrexate Placebo vs Methotrexate, 2.5 mg, Plus Abatacept Placebo; Test type: Superiority or Other; Odds Ratio (OR) = 2.04, 95% CI 2-sided [0.81 to 5.14], Standard Error of Mean 0.96 — At Months 12 and 18

3. Secondary Outcome: Percentage of Participants With Remission by Disease Activity Score 28 Based on C-reactive Protein (DAS28-CRP) Criteria Over Time - Intent to Treat Population
Description: TP=treatment period; WP=withdrawal period. Remission defined as DAS28-CRP<2.6. The DAS 28-CRP is a measure of disease activity in rheumatoid arthritis (RA) and assesses the 28 joints RA commonly affects; the score includes the number of tender and swollen joints (out of 28), CRP level (a measure of inflammation in the blood), and the patient's global assessment of health (ranging from very good to very bad). DAS-CRP scores range from 0 to 10, with higher values indicating greater disease activity. Individual measures are fed into a complex mathematical formula to produce the overall DAS (a score greater than 5.1 implies active disease; less than 3.2, well controlled disease; and less than 2.6, remission.)
Time Frame: Randomization to Month 24
Population: All randomized participants who received at least 1 dose of double-blind study medication in the Treatment Period. Percentage calculated as a/b, where a=number of patients who achieved remission at Day x, and b=number of patients in the analysis (intent to treat).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116 | 116
Percentage of participants
  TP Day 29 | 13.4 [7.32 to 19.57] | 8.6 [3.51 to 13.73] | 6.0 [1.70 to 10.37]
  TP Day 57 | 24.4 [16.66 to 32.08] | 11.2 [5.47 to 16.95] | 9.5 [4.15 to 14.81]
  TP Day 85 | 36.1 [27.50 to 44.77] | 21.6 [14.07 to 29.03] | 17.2 [10.37 to 24.12]
  TP Day 113 | 37.8 [29.10 to 46.53] | 29.3 [21.03 to 37.59] | 19.0 [11.83 to 26.10]
  TP Day 141 | 45.4 [36.43 to 54.32] | 29.3 [21.03 to 37.59] | 25.0 [17.12 to 32.88]
  TP Day 169 | 45.4 [36.43 to 54.32] | 32.8 [24.22 to 41.30] | 26.7 [18.67 to 34.78]
  TP Day 197 | 52.1 [43.13 to 61.08] | 36.2 [27.46 to 44.95] | 25.9 [17.89 to 33.83]
  TP Day 225 | 57.1 [48.25 to 66.03] | 40.5 [31.58 to 49.45] | 30.2 [21.82 to 38.53]
  TP Day 253 | 62.2 [53.47 to 70.90] | 37.9 [29.10 to 46.76] | 30.2 [21.82 to 38.53]
  TP 281 | 51.3 [42.28 to 60.24] | 42.2 [33.25 to 51.23] | 32.8 [24.22 to 41.30]
  TP 309 | 56.3 [47.39 to 65.21] | 37.9 [29.10 to 46.76] | 36.2 [27.46 to 44.95]
  TP Day 337 | 63.0 [54.35 to 71.70] | 43.1 [34.09 to 52.12] | 33.6 [25.02 to 42.22]
  TP 365 | 61.3 [52.60 to 70.09] | 43.1 [34.09 to 52.12] | 45.7 [36.62 to 54.75]
  WP Day 29 | 51.3 [42.28 to 60.24] | 36.2 [27.46 to 44.95] | 27.6 [19.45 to 35.72]
  WP Day 57 | 40.3 [31.52 to 49.15] | 25.0 [17.12 to 32.88] | 18.1 [11.10 to 25.11]
  WP Day 85 | 31.1 [22.78 to 39.41] | 18.1 [11.10 to 25.11] | 18.1 [11.10 to 25.11]
  WP Day 169 | 19.3 [12.23 to 26.42] | 12.9 [6.82 to 19.04] | 9.5 [4.15 to 14.81]
  WP Day 253 | 17.6 [10.80 to 24.50] | 9.5 [4.15 to 14.81] | 13.8 [7.52 to 20.07]
  WP Day 365 | 9.2 [4.04 to 14.45] | 6.0 [1.70 to 10.37] | 6.0 [1.70 to 10.37]

4. Secondary Outcome: Adjusted Mean Change From Baseline in Disease Activity Score 28 Based on C-reactive Protein (DAS28-CRP) at Months 6, 12, and 18
Description: TP=treatment period; WP=withdrawal period. The DAS 28-CRP is a measure of disease activity in rheumatoid arthritis (RA) that assesses the 28 joints RA commonly affects; the score includes the number of tender and swollen joints (out of 28), CRP level (a measure of inflammation in the blood), and the patient's global assessment of health (ranging from very good to very bad). DAS-CRP scores range from 0 to 10, with higher values indicating greater disease activity. Individual measures are fed into a complex mathematical formula to produce the overall DAS (a score greater than 5.1 implies active disease; less than 3.2, well controlled disease; and less than 2.6, remission.)
Time Frame: Baseline to Month 18
Population: All randomized participants who received at least 1 dose of double-blind study medication in the Treatment Period. n=number evaluable
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116 | 116
Units on a scale
  Month 6 (TP Day 169) (n=102, 96, 101) | -2.72 (0.12) | -2.33 (0.12) | -1.93 (0.12)
  Month 12 (TP Day 365) (n=95, 84, 91) | -3.09 (0.13) | -2.75 (0.13) | -2.58 (0.13)
  Month 18 (WP Day 169) (n=41, 31, 32) | -1.54 (0.26) | -1.51 (0.29) | -1.06 (0.29)

5. Secondary Outcome: Percentage of Participants Who Achieved Remission by Criteria of the Simplified Disease Activity Index (SDAI) at Months 12 and 18
Description: TP=treatment period; WP=withdrawal period. SDAI-defined remission= ≤3.3. The SDAI is the simple linear sum of 5 outcome parameters: tender joint count (TJC) and swollen joint count (SJC) (based on a 28-joint assessment); patient's and physician's global assessments of disease activity (assessed on 0-10 cm visual analog scale, on which higher scores=greater affection due to disease activity); and C-reactive protein level (mg/dL). SDAI total score=0-86. SDAI <=3.3 indicates disease remission, >3.4 to 11=low disease activity, >11 to 26=moderate disease activity, and >26=high disease activity. TJC is assessed and recorded at each visit, with no swelling=0, swelling=1. SJC is assessed through identification of joints that are painful under pressure or to passive motion. TJC is recorded on the joint assessment form at each visit, with no tenderness =0, tenderness = 1. Higher score indicates greater affection due to disease activity.
Time Frame: Randomization to Month 18
Population: All randomized participants who received at least 1 dose of double-blind study medication in the Treatment Period. Percentage calculated as a/b, where a=number of patients who achieved remission at Months 12 and 18, and b=number of patients in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116 | 116
Percentage of participants
  Month 12 (TP Day 365) | 42.0 [33.15 to 50.89] | 29.3 [21.03 to 37.59] | 25.0 [17.12 to 32.88]
  Month 18 (WP Day 169) | 10.9 [5.32 to 16.53] | 8.6 [3.51 to 13.73] | 6.9 [2.29 to 11.51]

6. Secondary Outcome: Adjusted Mean Change From Baseline in Scores on Simplified Disease Activity Index (SDAI) Over Time
Description: TP=treatment period; WP=withdrawal period. The SDAI is the simple linear sum of 5 outcome parameters: swollen joint count (SJC) and tender joint count (TJC) (based on a 28-joint assessment); patient's and physician's global assessments of disease activity (assessed on 0-10 cm visual analog scale, on which higher scores=greater affection due to disease activity); and C-reactive protein level (mg/dL). SDAI total score=0-86. SJC is assessed and recorded at each visit, with no swelling=0, swelling=1 (higher score indicates greater swelling). TJC is assessed at each visit through identification of joints that are painful under pressure or to passive motion, with no tenderness=0, tenderness=1 (higher score indicates greater affection due to disease activity)..
Time Frame: Randomization to Month 18
Population: Intent to Treat (ITT) population. n= number of participants with both post baseline and baseline measurements.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116 | 116
Units on a scale
  TP Day 29 (n=109, 101, 107) | -13.11 (1.33) | -12.14 (1.37) | -10.12 (1.33)
  TP Day 57 (n=108, 101, 103) | -18.90 (1.25) | -15.83 (1.28) | -15.99 (1.26)
  TP Day 85 (n=108, 99, 103) | -24.13 (1.16) | -20.51 (1.20) | -19.55 (1.17)
  TP Day 113 (n=103, 98, 101) | -25.47 (1.12) | -23.56 (1.15) | -21.02 (1.13)
  TP Day 141 (n=104, 96, 104) | -27.15 (1.10) | -25.99 (1.13) | -22.14 (1.10)
  TP Day 169 (n=102, 96, 100) | -28.42 (1.08) | -26.20 (1.11) | -22.80 (1.09)
  TP Day 197 (n=103, 97, 96) | -29.66 (1.01) | -27.57 (1.03) | -24.37 (1.02)
  TP Day 225 (n=99, 94, 92) | -30.13 (1.04) | -28.39 (1.06) | -24.73 (1.06)
  TP Day 253 (n=98, 94, 91) | -31.14 (1.04) | -28.10 (1.06) | -25.80 (1.05)
  TP 281 (n=96, 93, 89) | -30.98 (1.10) | -28.16 (1.12) | -26.23 (1.12)
  TP 309 (n=91, 87, 92) | -30.82 (1.16) | -27.79 (1.18) | -26.36 (1.17)
  TP Day 337 (n=93, 84, 87) | -31.11 (1.15) | -29.34 (1.19) | -27.26 (1.17)
  TP 365 (n=95, 84, 91) | -31.24 (1.17) | -28.88 (1.21) | -28.34 (1.19)
  WP Day 29 (n=73, 59, 64) | -30.42 (1.32) | -28.05 (1.39) | -23.52 (1.36)
  WP Day 57 (n=69, 54, 59) | -27.68 (1.59) | -24.17 (1.74) | -17.94 (1.68)
  WP Day 85 (n=67, 47, 52) | -22.00 (2.18) | -21.55 (2.57) | -17.54 (2.44)
  WP Day 169 (n=41, 31, 32) | -17.43 (2.82) | -19.13 (3.25) | -13.64 (3.19)

7. Secondary Outcome: Percentage of Participants Achieving a Health Assessment Questionnaire (HAQ) Response Over Time
Description: HAQ response defined as a reduction of at least 0.3 units from baseline in score on the Health Assessment Questionnaire Disability Index (HAQ-DI), which assesses patients' functional ability by rating their abilities over the previous week. The HAQ-DI includes at least 2 questions from each of 8 categories: dressing and grooming, hygiene, arising, reach, eating, grip, walking, and common daily activities. Patients rate difficulty performing specific tasks: 0=without difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The sum of the categories score (the highest scored item in the category) is divided by the number of categories answered, yielding a score from 0-3. When aids, devices, or help is indicated by the patient, the score for the category item is raised from a 0 or a 1 to a 2, but if the patient's highest score for a subcategory is a 3, it stays a 3.
Time Frame: Randomization to Month 24
Population: All randomized participants who received at least 1 dose of double-blind study medication in the Treatment Period. Percentage calculated as a/b, where a=number of patients who achieved remission at Day x, and b=number of patients in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116 | 116
Percentage of participants
  TP Day 29 | 42.0 [33.15 to 50.89] | 31.0 [22.62 to 39.45] | 21.6 [14.07 to 29.03]
  TP Day 57 | 55.5 [46.53 to 64.39] | 44.0 [34.93 to 53.00] | 37.9 [29.10 to 46.76]
  TP Day 85 | 63.0 [54.35 to 71.70] | 45.7 [36.62 to 54.75] | 41.4 [32.42 to 50.34]
  TP Day 113 | 63.0 [54.35 to 71.70] | 49.1 [40.04 to 58.24] | 45.7 [36.62 to 54.75]
  TP Day 141 | 62.2 [53.47 to 70.90] | 51.7 [42.63 to 60.82] | 44.0 [34.93 to 53.00]
  TP Day 169 | 63.9 [55.23 to 72.50] | 56.0 [47.00 to 65.07] | 41.4 [32.42 to 50.34]
  TP Day 197 | 66.4 [57.90 to 74.87] | 59.5 [50.55 to 68.42] | 41.4 [32.42 to 50.34]
  TP Day 225 | 66.4 [57.90 to 74.87] | 57.8 [48.77 to 66.75] | 38.8 [29.93 to 47.66]
  TP Day 253 | 68.9 [60.59 to 77.22] | 55.2 [46.12 to 64.22] | 45.7 [36.62 to 54.75]
  TP Day 281 | 64.7 [56.12 to 73.29] | 56.9 [47.88 to 65.91] | 46.6 [37.47 to 55.63]
  TP Day 309 | 65.5 [57.01 to 74.08] | 56.9 [47.88 to 65.91] | 46.6 [37.47 to 55.63]
  TP Day 337 | 64.7 [56.12 to 73.29] | 55.2 [46.12 to 64.22] | 46.6 [37.47 to 55.63]
  TP Day 365 | 67.2 [58.79 to 75.66] | 52.6 [43.50 to 61.67] | 44.0 [34.93 to 53.00]
  WP Day 29 | 52.1 [43.13 to 61.08] | 39.7 [30.75 to 48.56] | 37.1 [28.28 to 45.86]
  WP Day 57 | 43.7 [34.79 to 52.61] | 34.5 [25.83 to 43.13] | 26.7 [18.67 to 34.78]
  WP Day 85 | 39.5 [30.71 to 48.28] | 28.4 [20.24 to 36.66] | 23.3 [15.59 to 30.97]
  WP Day 169 | 22.7 [15.16 to 30.21] | 16.4 [9.64 to 23.11] | 10.3 [4.80 to 15.89]
  WP Day 253 | 15.1 [8.69 to 21.56] | 9.5 [4.15 to 14.81] | 6.9 [2.29 to 11.51]
  WP Day 365 | 10.1 [4.67 to 15.49] | 6.9 [2.29 to 11.51] | 5.2 [1.14 to 9.20]

8. Secondary Outcome: Adjusted Mean Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Over Time
Description: The Health Assessment Questionnaire Disability Index (HAQ-DI) assesses patients' functional ability by rating their abilities over the previous week. The HAQ-DI includes at least 2 questions from each of 8 categories: dressing and grooming, hygiene, arising, reach, eating, grip, walking, and common daily activities. Patients rate difficulty performing specific tasks: 0=without difficulty, 1=with some difficulty, 2=with much difficulty, and 3=unable to do. The sum of the categories score (the highest scored item in the category) is divided by the number of categories answered, yielding a score from 0-3. When aids, devices, or help is indicated by the patient, the score for the category item is raised from a 0 or a 1 to a 2, but if the patient's highest score for a subcategory is a 3, it stays a 3.
Time Frame: Randomization to Month 18
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116 | 116
Units on a scale
  TP Day 29 (n=104, 103, 91) | -0.33 (0.05) | -0.21 (0.05) | -0.09 (0.05)
  TP Day 57 (n=102, 100, 93) | -0.48 (0.05) | -0.38 (0.05) | -0.32 (0.05)
  TP Day 85 (n=105, 97, 88) | -0.64 (0.05) | -0.45 (0.05) | -0.40 (0.05)
  TP Day 113 (n=105, 98, 90) | -0.67 (0.05) | -0.55 (0.05) | -0.50 (0.05)
  TP Day 141 (n=100, 98, 88) | -0.72 (0.05) | -0.53 (0.05) | -0.46 (0.06)
  TP Day 169 (n=95, 95, 85) | -0.74 (0.05) | -0.59 (0.05) | -0.52 (0.06)
  TP Day 197 (n=99, 96, 83) | -0.78 (0.05) | -0.62 (0.06) | -0.54 (0.06)
  TP Day 225 (n=98, 95, 83) | -0.79 (0.06) | -0.67 (0.06) | -0.56 (0.06)
  TP Day 253 (n=96, 91, 84) | -0.82 (0.05) | -0.65 (0.06) | -0.63 (0.06)
  TP Day 281 (n=90, 93, 81) | -0.82 (0.06) | -0.65 (0.06) | -0.62 (0.06)
  TP Day 309 (n=89, 88, 82) | -0.81 (0.06) | -0.67 (0.06) | -0.66 (0.06)
  TP Day 337 (n=88, 85, 80) | -0.84 (0.06) | -0.70 (0.06) | -0.70 (0.06)
  TP Day 365 (n=90, 82, 77) | -0.87 (0.06) | -0.73 (0.06) | -0.72 (0.06)
  WP Day 29 (n=70, 55, 55) | -0.85 (0.06) | -0.67 (0.07) | -0.63 (0.07)
  WP Day 57 (n=66, 53, 54) | -0.67 (0.07) | -0.58 (0.08) | -0.39 (0.08)
  WP Day 85 (n=65, 45, 46) | -0.54 (0.08) | -0.48 (0.09) | -0.37 (0.09)
  WP Day 169 (n=34, 28, 26) | -0.52 (0.10) | -0.49 (0.11) | -0.33 (0.12)

9. Secondary Outcome: Adjusted Mean Change From Baseline at Months 6, 12, and 18 in Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores of Short Form-36 (SF-36)
Description: TP=treatment period; WP=withdrawal period. The SF-36 is a 36-item self-administered questionnaire developed to assess health-related quality of life (QOL) and comprises 8 domains, including 4 physical (physical health, bodily pain, physical functioning and physical role limitations) and 4 mental (mental health, vitality, social functioning, and emotional role limitation) subscales. Responses are used to derive physical and mental component summary scores, ranging from 0 to 100, with higher scores indicating better QOL (0=Poorest Health; 100=Best Health). Mean change from baseline=postbaseline value-baseline value; a higher value signifies improvement.
Time Frame: Randomization to Months 6, 12, and 18
Population: as for outcome 4
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116 | 116
Units on a scale
  PCS score TP Day 169 (n=106, 95, 96) | 11.68 (0.82) | 9.16 (0.86) | 7.47 (0.85)
  PCS score TP Day 365 (n=94, 88, 91) | 13.91 (0.93) | 10.23 (0.97) | 10.92 (0.95)
  PCS score WP Day 169 (n=48, 36, 37) | 6.16 (1.45) | 4.59 (1.65) | 6.27 (1.63)
  MCS score TP Day 169 (n=106, 95, 96) | 6.11 (0.92) | 3.99 (0.97) | 4.69 (0.95)
  MCS score TP Day 365 (n=94, 88, 91) | 7.67 (1.04) | 5.48 (1.08) | 7.23 (1.06)
  MCS score WP Day 169 (n=48, 36, 37) | 2.75 (1.44) | 4.36 (1.64) | 2.23 (1.63)

10. Secondary Outcome: Adjusted Mean Change From Baseline Over Time in Findings on Magnetic Resonance Imaging (MRI)
Description: TP=treatment period; WP=withdrawal period. Change from Baseline=Postbaseline-baseline value. MRI was used to assess joint damage progression at Months 6, 12, and 18. If >20% of joints with a missing score for a parameter (erosion, osteitis, and synovitis), the MRI score of each parameter was considered missing. If ≤20% of joints had a missing score for a parameter, the MRI score for that parameter from the missing joints was carried forward from the previous MRI assessment, or carried backward from the next MRI assessment, if missing score occurred at baseline. MRI total score ranged from 0 (best outcome) to 4 (worst outcome). A gadolinium-enhanced MRI of the dominant hand-wrist was performed on all randomized patients at 5 points. The hand/wrist assessed to have more synovitis was selected initially and used for all subsequent evaluations. The MRI examination was standardized to ensure sufficient image quality for the evaluation of radiographic progression of rheumatoid arthritis.
Time Frame: Randomization to Month 18
Population: All randomized participants who received at least 1 dose of double-blind study medication in the Treatment Period. n=the number of patients with both baseline and postbaseline measurements.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116 | 116
Units on a scale
  Osteitis TP Day 169 (n=93, 94, 89) | -2.03 (0.47) | -1.13 (0.47) | -0.73 (0.48)
  Osteitis TP Day 365 (n=83, 74, 78) | -2.32 (0.46) | -1.30 (0.46) | -0.90 (0.46)
  Osteitis WP Day 169 (n=31, 30, 25) | -1.94 (0.88) | 0.98 (0.89) | -0.33 (0.96)
  Erosion TP Day 169 (n=93, 94, 89) | 0.26 (0.28) | 1.15 (0.28) | 1.15 (0.28)
  Erosion TP Day 365 (n=83, 74, 78) | 0.34 (0.35) | 1.57 (0.36) | 1.56 (0.36)
  Erosion WP Day 169 (n=31, 30, 25) | 0.20 (0.47) | 2.16 (0.48) | 1.89 (0.50)
  Synovitis TP Day 169 (n=93, 94, 89) | -1.82 (0.21) | -0.93 (0.21) | -0.78 (0.21)
  Synovitis TP Day 365 (n=83, 74, 78) | -2.38 (0.29) | -1.36 (0.30) | -0.77 (0.30)
  Synovitis WP Day 169 (n=31, 30, 25)) | -1.71 (0.45) | -0.95 (0.45) | -0.71 (0.49)

11. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Related SAEs, Discontinuations Due to SAEs, Related Adverse Events (AEs), and Discontinuations Due to AEs During the Treatment Period
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=having certain, probable, possible, or unknown relationship to study drug.
Time Frame: Day 1 to up to 56 days following the last dosing day (Day 365); all deaths during study period, including those that occurred >56 days after last dose in Treatment Period
Population: All randomized participants who received at least 1 dose of double-blind study medication in the Treatment Period
Measure: Number; unit: Participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116 | 116
Participants
  Deaths | 0 | 0 | 2
  SAEs | 8 | 14 | 9
  Related SAEs | 3 | 3 | 1
  Discontinuations due to SAEs | 2 | 5 | 3
  Related AEs | 53 | 48 | 51
  Discontinuations due to AEs | 4 | 8 | 5

12. Secondary Outcome: Adverse Events (AEs) of Interest During the Treatment Period
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=having certain, probable, possible, or unknown relationship to study drug. AEs of special interest are events potentially associated with the drug or disease under study.
Time Frame: Day 1 to 56 days following last dosing day (Day 365)
Population: All randomized participants who received at least 1 dose of double-blind study medication in the Treatment Period
Measure: Number; unit: Participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116 | 116
Participants
  Infections | 68 | 64 | 69
  Malignancy | 1 | 2 | 1
  Autoimmune disorders (prespecified) | 1 | 2 | 3
  Local injection site reactions (prespecified) | 2 | 0 | 0

13. Secondary Outcome: Number of Participants With Results on Hematology and Clinical Laboratory Tests Meeting the Criteria for Marked Abnormality During Treatment Period
Description: Lower limit of normal (LLN); Upper limit of normal (ULN); Pretreatment (preRX). Criteria for marked abnormality: Platelet count (*10^9 c/µL) <0.67*LLN or >1.5*ULN, or if preRX<LLN, use 0.5*preRX and <100,000/mm^3; potassium, serum (mEq) <0.9*LLN or >1.1*ULN, or if preRX <LLN, use <0.9*preRX or >ULN if preRX>ULN, use >1.1*preRX or <LLN; blood urea nitrogen (mg/dL) >2*preRX; creatinine (mg/dL) >1.5*preRX; ALT (U/L) >3*ULN, or if preRX>ULN, use >4*preRX; AST (U/L) >3*ULN, or if preRX>ULN, use >4*preRX; ALP (U/L) >2*ULN, or if preRX>ULN, use >3*preRX; G-glutamyl transferase U/L) >2*ULN, or if preRX>ULN, use >3*preRX; glucose, fasting (mg/dL) <0.8*LLN or >1.5*ULN, or if preRX<LLN use <0.8*preRX or >ULN if preRX >ULN, use >2.0*preRX or OR <LLN; glucose, serum (mg/dL) <65 or >220; uric acid (mg/dL)>1.5*ULN, or if preRX, use >2*preRX; albumin (g/dL) <0.9*LLN, or if preRX<LLN, use <0.75*preRX; hemoglobin (g/dL)>3 decrease from preRX; hematocrit (%) < 0.75*preRX.
Time Frame: Day 1 up to 56 days following the last dosing day in the Treatment Period (Day 365)
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116 | 116
Participants
  Platelet count (high) (n=119, 116, 115) | 2 | 0 | 0
  Potassium, serum (low) | 1 | 1 | 1
  Blood urea nitrogen (high) | 4 | 1 | 2
  Creatinine (high) | 2 | 1 | 3
  Alanine aminotransferase (ALT)(high) | 3 | 0 | 2
  Aspartate aminotransferase (AST)(high) | 2 | 0 | 1
  G-glutamyl transferase (GGT) (high) | 3 | 1 | 1
  Glucose, fasting (low) (n=78, 72, 75) | 2 | 0 | 2
  Glucose, fasting (high) (n=78, 72, 75) | 1 | 2 | 1
  Glucose, serum (low) (n=84, 78, 75) | 5 | 6 | 2
  Glucose, serum (high) (n=84, 78, 75) | 1 | 4 | 3
  Uric acid (high) | 0 | 1 | 0
  Albumin (low) | 1 | 1 | 4
  Hemoglobin (low) (n=119, 116, 115) | 0 | 2 | 0
  Hematocrit (low) (n=119, 116, 115) | 0 | 2 | 0

14. Secondary Outcome: Percentage of Participants With Remission by Disease Activity Score 28 Based on C-reactive Protein (DAS28-CRP) Criteria Over Time During Withdrawal Period- Treated Participants in Remission at Month 12
Description: WP=withdrawal period. Remission defined as DAS28-CRP<2.6. The DAS 28-CRP is a measure of disease activity in rheumatoid arthritis (RA) and assesses the 28 joints RA commonly affects; the score includes the number of tender and swollen joints (out of 28), CRP level (a measure of inflammation in the blood), and the patient's global assessment of health (ranging from very good to very bad). DAS-CRP scores range from 0 to 10, with higher values indicating greater disease activity. Individual measures are fed into a complex mathematical formula to produce the overall DAS (a score greater than 5.1 implies active disease; less than 3.2, well controlled disease; and less than 2.6, remission.). Percentage= number of participants with remission divided by number of participants who were analyzed (all treated participants who were in remission at end of treatment period and entered the Withdrawal Period)
Time Frame: End of Treatment Period (Month 12) to End of Withdrawal Period (Month 24)
Population: Treated participants who were in remission at Month 12 (DAS28-CRP<2.6) and entered the Withdrawal Period were analyzed.( N=number of participants analyzed).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Abatacept, 125 mg, Plus Methotrexate, 2.5 mg: Participants received abatacept, 125 mg subcutaneously, plus methotrexate (MTX), 2.5 mg orally as tablets, once weekly, during the 12-month Treatment Period. Participants with a Low Disease Activity Score (LDAS) defined as DAS28-CRP score of < 3.2 at Month 12 (end of Treatment Period) entered the Withdrawal Period for up to 12 months, during which all study medication was withdrawn. Participants with a DAS28-CRP score of >3.2 were discontinued from the study. All MTX and corticosteroids, if not already discontinued, were to be tapered off during the first month of the Withdrawal Period. Participants who experienced a worsening of rheumatoid arthritis (RA) symptoms or a RA flare after at least 3 months in the Withdrawal Period were eligible to enroll into a 6-month Re-exposure Period, during which they received open-label treatment with abatacept SC (125 mg/week) and MTX.
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 73 | 50 | 53
percentage of participants
  WP Day 29 | 73.3 [65.46 to 85.23] | 72.0 [59.55 to 84.45] | 54.7 [41.32 to 68.12]
  WP Day 57 | 58.9 [47.62 to 70.19] | 56.0 [42.24 to 69.76] | 32.1 [19.51 to 44.64]
  WP Day 85 | 42.5 [31.13 to 53.80] | 40.0 [26.42 to 53.58] | 35.8 [22.94 to 48.76]
  WP Day 169 | 26.0 [15.96 to 36.09] | 30.0 [17.30 to 42.70] | 17.0 [6.87 to 27.09]
  WP Day 253 | 20.5 [11.28 to 29.82] | 22.0 [10.52 to 33.48] | 20.8 [9.84 to 31.67]
  WP Day 365 | 12.3 [4.79 to 19.87] | 14.0 [4.38 to 23.62] | 11.3 [2.79 to 19.85]

15. Secondary Outcome: Percentage of Participants Who Achieved Remission by Criteria of the Simplified Disease Activity Index (SDAI) Over Time in Treatment Period and Withdrawal Period
Description: TP=treatment period; WP=withdrawal period. SDAI-defined remission= ≤3.3. The SDAI is the simple linear sum of 5 outcome parameters: tender joint count (TJC) and swollen joint count (SJC) (based on a 28-joint assessment); patient's and physician's global assessments of disease activity (assessed on 0-10 cm visual analog scale, on which higher scores=greater affection due to disease activity); and C-reactive protein level (mg/dL). SDAI total score=0-86. SDAI <=3.3 indicates disease remission, >3.4 to 11=low disease activity, >11 to 26=moderate disease activity, and >26=high disease activity. TJC is assessed and recorded at each visit, with no swelling=0, swelling=1. SJC is assessed through identification of joints that are painful under pressure or to passive motion. TJC is recorded on the joint assessment form at each visit, with no tenderness =0, tenderness = 1. Higher score indicates greater affection due to disease activity. Percent=number with remission/number evaluated (ITT)
Time Frame: Randomization to Month 24
Population: ITT analysis population: Included all randomized participants who received at least 1 dose of double-blind study medication in the Treatment Period. Participants were grouped according to the treatment regimen to which they were randomized.N= number evaluated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116 | 116
percentage of participants
  TP Day 29 | 4.2 [1.38 to 9.53] | 3.4 [0.95 to 8.59] | 1.7 [0.21 to 6.09]
  TP Day 57 | 9.2 [4.71 to 15.94] | 6.0 [2.46 to 12.04] | 1.7 [0.21 to 6.09]
  TP Day 85 | 17.6 [10.80 to 24.50] | 8.6 [3.51 to 13.73] | 6.0 [1.70 to 10.37]
  TP Day 113 | 23.5 [15.91 to 31.15] | 17.2 [10.37 to 24.12] | 7.8 [2.89 to 12.63]
  TP Day 141 | 31.9 [23.56 to 40.31] | 23.3 [15.59 to 30.97] | 10.3 [4.80 to 15.89]
  TP Day 169 | 31.1 [22.78 to 39.41] | 20.7 [13.32 to 28.06] | 11.2 [5.47 to 16.95]
  TP Day 197 | 33.6 [25.13 to 42.10] | 21.6 [14.07 to 29.03] | 12.9 [6.82 to 19.04]
  TP Day 225 | 38.7 [29.91 to 47.40] | 25.9 [17.89 to 33.83] | 14.7 [8.22 to 21.09]
  TP Day 253 | 37.8 [29.10 to 46.53] | 25.0 [17.12 to 32.88] | 13.8 [7.52 to 20.07]
  TP Day 281 | 37.8 [29.10 to 46.53] | 26.7 [18.67 to 34.78] | 18.1 [11.10 to 25.11]
  TP Day 309 | 40.3 [31.52 to 49.15] | 26.7 [18.67 to 34.78] | 19.0 [11.83 to 26.10]
  TP Day 337 | 41.2 [32.33 to 50.02] | 31.0 [22.62 to 39.45] | 19.0 [11.83 to 26.10]
  TP Day 365 | 42.0 [33.15 to 50.89] | 29.3 [21.03 to 37.59] | 25.0 [17.12 to 32.88]
  WP Day 29 | 38.7 [29.91 to 47.40] | 26.7 [18.67 to 34.78] | 14.7 [8.22 to 21.09]
  WP Day 57 | 26.9 [18.92 to 34.86] | 20.7 [13.32 to 28.06] | 10.3 [4.80 to 15.89]
  WP Day 85 | 21.0 [13.69 to 28.33] | 15.5 [8.93 to 22.11] | 14.7 [8.22 to 21.09]
  WP Day 169 | 11.8 [5.98 to 17.55] | 9.5 [4.15 to 14.81] | 6.9 [2.29 to 11.51]
  WP Day 253 | 11.8 [5.98 to 17.55] | 9.5 [4.15 to 14.81] | 7.8 [2.89 to 12.63]
  WP Day 365 | 6.7 [2.22 to 11.22] | 4.3 [0.61 to 8.01] | 4.3 [0.61 to 8.01]

16. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs) and Discontinuations Due to AEs During the Full Study (All Periods)
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Includes data up to last active dose date +56 days if the participant discontinued the Treatment Period or did not enter the Withdrawal Period, up to the day of discontinuation in the Withdrawal Period for participants discontinuing the Withdrawal Period without entering the Re-exposure Period (RP), up to Day 729 visit (Month 24) for participants who complete the Withdrawal Period, and up to 56 days post last active dose in Re-exposure Period for participants entering the Re-exposure Period.
Time Frame: Day 1 to 56 days post last dose in the study, up to Month 30
Population: All randomized participants who received at least 1 dose of study medication were analyzed.
Measure: Number; unit: participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 119 | 116 | 116
participants
  Death | 0 | 0 | 2
  SAE | 11 | 15 | 15
  Discontinued Due to AE | 4 | 8 | 7

17. Secondary Outcome: Adverse Events (AEs) of Interest During the Withdrawal Period
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. AEs of special interest are events potentially associated with the drug or disease under study. Includes events with an onset date on or after 57 days post last dosing day (active abatacept or active MTX whichever is the later) in the Treatment Period and up to end of Withdrawal Period. Treatment groups represent treatment received during the Treatment Period.
Time Frame: Last dose in TP + 57 days, up to Month 24
Population: All randomized participants who received at least 1 dose of double-blind study medication in the Treatment Period and entered the Withdrawal Period. Treatment groups represent treatment during the TP.
Measure: Number; unit: participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 84 | 66 | 75
participants
  Infections | 8 | 6 | 10
  Malignancy | 1 | 0 | 1
  Autoimmune disorders (prespecified) | 0 | 0 | 1
  Local injection site reactions(prespecified) | 0 | 0 | 0

18. Secondary Outcome: Adverse Events (AEs) of Interest During the Re-exposure Period
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. AEs of special interest are events potentially associated with the drug or disease under study. Includes data up to 56 days post the last dosing day (active abatacept or active MTX, whichever is the later) in the Re-exposure Period. Treatment groups represent Treatment received during Treatment Period.
Time Frame: First dose in Re-exposure period up to last dose of Re-exposure Period + 56 days
Population: Includes data up to 56 days post the last dosing day (active abatacept or active MTX, whichever is the later) in the Re-exposure Period. Treatment groups represent Treatment received during Treatment Period.
Measure: Number; unit: participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 55 | 48 | 43
participants
  Infections | 17 | 8 | 12
  Malignancy | 0 | 0 | 0
  Autoimmune Disorders (prespecified) | 0 | 0 | 0
  Local Injection site reactions (prespecified) | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Results on Hematology and Clinical Laboratory Tests Meeting the Criteria for Marked Abnormality in Withdrawal Period
Description: LLN=lower limit of normal; ULN=upper limit of normal; preRX=pretreatment. Criteria for marked abnormality on laboratory test results: Platelet count (*10^9 c/µL) <0.67*LLN or >1.5*ULN, or if preRX<LLN, use 0.5*preRX and <100,000/mm^3; potassium, serum (mEq) <0.9*LLN or >1.1*ULN, or if preRX <LLN, use <0.9*preRX or >ULN if preRX>ULN, use >1.1*preRX or <LLN; blood urea nitrogen (mg/dL) >2*preRX; creatinine (mg/dL) >1.5*preRX; ALT (U/L) >3*ULN, or if preRX>ULN, use >4*preRX; AST (U/L) >3*ULN, or if preRX>ULN, use >4*preRX; ALP (U/L) >2*ULN, or if preRX>ULN, use >3*preRX; G-glutamyl transferase (GGT) (U/L) >2*ULN, or if preRX>ULN, use >3*preRX; glucose, fasting (mg/dL) <0.8*LLN or >1.5*ULN, or if preRX<LLN use <0.8*preRX or >ULN if preRX >ULN, use >2.0*preRX or OR <LLN; glucose, serum (mg/dL) <65 or >220; uric acid (mg/dL)>1.5*ULN, or if preRX, use >2*preRX; albumin (g/dL) <0.9*LLN, or if preRX<LLN, use <0.75*preRX; hemoglobin (g/dL)>3 decrease from preRX; hematocrit (%) < 0.75*preRX.
Time Frame: Last dose in TP + 57 days, up to Month 24
Population: All randomized participants who received at least 1 dose of study drug in the Treatment Period, entered the Withdrawal Period, and had values available. n=number evaluable
Measure: Number; unit: participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 60 | 52 | 48
participants
  Hemoglobin Low (n=60, 52, 48) | 1 | 2 | 0
  Creatinine High (n=60, 52, 48) | 1 | 2 | 2
  Alanine aminotransferase (ALT) High (n=60, 52, 48) | 1 | 0 | 0
  GGT High (n=60, 52, 48) | 1 | 0 | 0
  Fasting Glucose High (30, 28, 25) | 0 | 2 | 1
  Glucose Low (n=36,31,27) | 5 | 3 | 0
  Glucose High (n=36, 31, 27) | 0 | 1 | 1

20. Secondary Outcome: Number of Participants With Results on Hematology and Clinical Laboratory Tests Meeting the Criteria for Marked Abnormality in Re-exposure Period
Description: LLN=lower limit of normal; ULN=upper limit of normal; preRX=pretreatment. Criteria for marked abnormality on laboratory test results: Platelet count (*10^9 c/µL) <0.67*LLN or >1.5*ULN, or if preRX<LLN, use 0.5*preRX and <100,000/mm^3; potassium, serum (mEq) <0.9*LLN or >1.1*ULN, or if preRX <LLN, use <0.9*preRX or >ULN if preRX>ULN, use >1.1*preRX or <LLN; blood urea nitrogen (mg/dL) >2*preRX; creatinine (mg/dL) >1.5*preRX; ALT (U/L) >3*ULN, or if preRX>ULN, use >4*preRX; AST (U/L) >3*ULN, or if preRX>ULN, use >4*preRX; ALP (U/L) >2*ULN, or if preRX>ULN, use >3*preRX; G-glutamyl transferase U/L) >2*ULN, or if preRX>ULN, use >3*preRX; glucose, fasting (mg/dL) <0.8*LLN or >1.5*ULN, or if preRX<LLN use <0.8*preRX or >ULN if preRX >ULN, use >2.0*preRX or OR <LLN; glucose, serum (mg/dL) <65 or >220; uric acid (mg/dL)>1.5*ULN, or if preRX, use >2*preRX; albumin (g/dL) <0.9*LLN, or if preRX<LLN, use <0.75*preRX; hemoglobin (g/dL)>3 decrease from preRX; hematocrit (%) < 0.75*preRX.
Time Frame: Start of re-exposure period to 56 days post last dose, up to Month 30
Population: All treated participants entering the Re-exposure Period and having measurements available were analyzed. n=evaluable. Treatment groups represent Treatment received during Treatment Period.
Measure: Number; unit: participants
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Number analyzed (Participants) | 55 | 48 | 43
participants
  Hematocrit Low (n=55,47,43) | 0 | 1 | 0
  Hemoglobin Low (n=55,48, 43) | 0 | 2 | 0
  Creatinine High (n=55, 48, 43) | 0 | 1 | 0
  ALT High (n=55, 48, 43) | 2 | 0 | 2
  ALP High (n=55, 48, 43) | 1 | 0 | 0
  AST High (n=55, 48, 43) | 2 | 0 | 1
  GGT High (n=55, 48, 43) | 2 | 0 | 1
  Fasting Glucose Low (n=33, 32, 28) | 1 | 0 | 0
  Fasting Glucose High (n=33, 32, 28) | 0 | 2 | 1
  Glucose Low (n=27,24,18) | 0 | 2 | 0
  Glucose High (n=27,24,18) | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Abatacept, 125 mg, Plus Methotrexate, 2.5 mg: Participants received abatacept, 125 mg subcutaneously, plus methotrexate, 2.5 mg orally as tablets, once weekly, during the 12-month Treatment Period. Participants with a LDAS defined as DAS28-CRP score of < 3.2 at Month 12 (end of Treatment Period) entered the Withdrawal Period for up to 12 months, during which all study medication was withdrawn. Participants with a DAS28-CRP score of >3.2 were discontinued from the study. All MTX and corticosteroids, if not already discontinued, were to be tapered off during the first month of the Withdrawal Period. Participants who experienced a worsening of RA symptoms or a RA flare after at least 3 months in the Withdrawal Period were eligible to enroll into a 6-month Re-exposure Period, during which they received open-label treatment with abatacept SC 125 mg/week and MTX. Safety data was collected from Day 1 to 56 days post last dose.
- Abatacept, 125 mg, Plus Methotrexate Placebo: Participants received abatacept, 125 mg subcutaneously, plus methotrexate placebo tablets orally, once weekly during the 12-month Treatment Period. Participants with a LDAS defined as DAS28-CRP score of < 3.2 at Month 12 (end of Treatment Period) entered the Withdrawal Period for up to 12 months, during which all study medication was withdrawn. Participants with a DAS28-CRP score of >3.2 were discontinued from the study. Participants who experienced a worsening of RA symptoms or a RA flare after at least 3 months in the Withdrawal Period were eligible to enroll into a 6-month Re-exposure Period, during which they received open-label treatment with abatacept SC (125 mg/week) and MTX. Safety data was collected from Day 1 to 56 days post last dose.
- Methotrexate, 2.5 mg, Plus Abatacept Placebo: Participants received methotrexate, 2.5 mg, orally as tablets, plus abatacept placebo subcutaneously, once weekly during the 12-month Treatment Period. Participants with a LDAS defined as DAS28-CRP score of < 3.2 at Month 12 (end of Treatment Period) entered the Withdrawal Period for up to 12 months, during which all study medication was withdrawn. Participants with a DAS28-CRP score of >3.2 were discontinued from the study. All MTX and corticosteroids, if not already discontinued, were to be tapered off during the first month of the Withdrawal Period. Participants who experienced a worsening of RA symptoms or a RA flare after at least 3 months in the Withdrawal Period were eligible to enroll into a 6-month Re-exposure Period, during which they received open-label treatment with abatacept SC (125 mg/week) and MTX. Safety data was collected from Day 1 to 56 days post last dose.
Arm/Group | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg | Abatacept, 125 mg, Plus Methotrexate Placebo | Methotrexate, 2.5 mg, Plus Abatacept Placebo
Serious Adverse Events (participants affected / at risk) | 11/119 | 15/116 | 15/116
Other Adverse Events (participants affected / at risk) | 81/119 | 64/116 | 78/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg (N=119) | Abatacept, 125 mg, Plus Methotrexate Placebo (N=116) | Methotrexate, 2.5 mg, Plus Abatacept Placebo (N=116)
Carotid artery occlusion (Nervous system disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Endometrial disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 3 | 1 | 2
Strangulated hernia (General disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Myocarditis post infection (Cardiac disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept, 125 mg, Plus Methotrexate, 2.5 mg (N=119) | Abatacept, 125 mg, Plus Methotrexate Placebo (N=116) | Methotrexate, 2.5 mg, Plus Abatacept Placebo (N=116)
Headache (Nervous system disorders) | 8 | 8 | 7
Pharyngitis (Infections and infestations) | 3 | 6 | 7
Urinary tract infection (Infections and infestations) | 14 | 15 | 15
Gastritis (Gastrointestinal disorders) | 4 | 1 | 7
Nausea (Gastrointestinal disorders) | 18 | 8 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 9 | 7
Mouth ulceration (Gastrointestinal disorders) | 6 | 5 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 1 | 1
Hypertension (Vascular disorders) | 4 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 5 | 8 | 4
Influenza (Infections and infestations) | 5 | 9 | 6
Sinusitis (Infections and infestations) | 9 | 4 | 2
Gastroenteritis (Infections and infestations) | 6 | 3 | 8
Nasopharyngitis (Infections and infestations) | 28 | 20 | 22
Abdominal pain upper (Gastrointestinal disorders) | 5 | 6 | 6
Bronchitis (Infections and infestations) | 8 | 6 | 10
Upper respiratory tract infection (Infections and infestations) | 15 | 15 | 20
Vomiting (Gastrointestinal disorders) | 6 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.